CLINICAL TRIAL: NCT00036166
Title: An Open-Label, Non-Comparative Study of FK463 for the Treatment of Invasive Aspergillosis
Brief Title: Study of FK463 for the Treatment of Invasive Aspergillosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FG463-21-01; 98-0-046 (Other: Alternate Protocol Number)
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2015-06

CONDITIONS: Aspergillosis
Keywords: Aspergillus; Anti-Fungal
MeSH Terms: conditions — Aspergillosis | interventions — Micafungin

INTERVENTIONS:
Drug: FK463

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of FK463 in patients with proven or probable invasive infections due to Aspergillus species.

DETAILED DESCRIPTION:
This will be an open-label, non-comparative study of intravenous FK463. Enrollment will include at least 100 patients evaluable for efficacy.

ELIGIBILITY:
Inclusion Criteria

* Has proven or probable systemic infection with Aspergillus species

Exclusion Criteria

* Has abnormal liver test parameters, e.g., AST or ALT > 10 times upper limit of normal
* Has bronchopulmonary aspergillosis, aspergillomas, sinus aspergillosis or external otitis but does not have histologic evidence of tissue invasion
* Has life-expectancy judged to be less than 5 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 1999-01-29 (Actual); Primary Completion 2002-01-31 (Actual); Study Completion 2002-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- Austria (2):
  - Medizinische Univ.-Klinik, Graz
  - Krankenhaus Elisabethinen Linz, Linz
- France (4):
  - Hopital Henri Mondor, Service d'Hematologie Clinique, Créteil
  - Hotel Dieu, Service d'Hematologie, Nantes
  - Hopital Saint Louis, Service D'Hematologie/Greffe de Moelle, Paris
  - Hopital Necker Enfants Malades, Service d'Hematologie, Paris
- Germany (7):
  - Johann Wolfgang Goethe Universitat, Medizinische Klinik III, Frankfurt
  - Westpfalz Krankehaus, Kaiserslautern
  - Medizinische Klinik und Poliklinik II, Abt. Hamatologie und Onkologie, Leipzig
  - Klinikum der Stadt, Medizinische Klinik A, Ludwigshafen
  - Uniklinik Mainz, Mainz
  - LMU Munchen, Hamatopoetische Zell - Transplantation, München
  - Universitat Wurzburg, Institut fur Molekulare und Infectionsbiologie, Würzburg
- Italy (2):
  - Nationale Institute for Cancer Research, Genova
  - Ospedale Niguarda-Ca Granda, Dept. of Internal Medicine Padiglione Brera, Milan
- Institute of Haematology and Blood Transfusion, Warsaw, Poland
- Spain (3):
  - Hospital Clinic I provencial, Servicio Enfermadades Infecciosas, Barcelona
  - Hospital Gregorio Maranon, Servicio de Enfermadades Infecciosas, Madrid
  - Hospital Doce de Octubre, Servicio de Microbiologia y Enfermadades Infecciosas, Madrid
- Huddinge University Hospital, Dept. of Transplantation Surgery/Immunology, Huddinge, Sweden
- United Kingdom (3):
  - Royal Free Hospital, Dept. of Haematological Oncology, London
  - Christie Hospital NHS Trust, Manchester
  - Royal Marsden Hospital, Sutton Surrey

REFERENCES:
- [Result] Denning DW, Marr KA, Lau WM, Facklam DP, Ratanatharathorn V, Becker C, Ullmann AJ, Seibel NL, Flynn PM, van Burik JA, Buell DN, Patterson TF. Micafungin (FK463), alone or in combination with other systemic antifungal agents, for the treatment of acute invasive aspergillosis. J Infect. 2006 Nov;53(5):337-49. doi: 10.1016/j.jinf.2006.03.003. Epub 2006 May 6. PMID 16678903
- [Result] Kontoyiannis DP, Ratanatharathorn V, Young JA, Raymond J, Laverdiere M, Denning DW, Patterson TF, Facklam D, Kovanda L, Arnold L, Lau W, Buell D, Marr KA. Micafungin alone or in combination with other systemic antifungal therapies in hematopoietic stem cell transplant recipients with invasive aspergillosis. Transpl Infect Dis. 2009 Feb;11(1):89-93. doi: 10.1111/j.1399-3062.2008.00349.x. Epub 2008 Oct 8. PMID 18983417
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=59